CLINICAL TRIAL: NCT02067351
Title: Mindfulness-Based Intervention in Breast Cancer Patients Undergoing Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniela L. Stan, M.D, Daniela Stan, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-008531
Record Dates: First submitted 2014-02-15; First posted 2014-02-20 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness Intervention (Experimental): Mindfulness intervention
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Meditation, body scan, yoga.

SUMMARY:
There is evidence that mindfulness-based interventions (MBIs) such as meditation, mindfulness-based stress reduction (MBSR) and yoga might improve Quality of Life (QOL) and reduce stress in breast cancer survivors. These interventions are becoming increasingly popular in cancer survivors. However, little is known about the feasibility and effect of MBIs administered during the interval of time of chemotherapy, on QOL and stress. The investigators are planning a MBI intervention study developed specifically for breast cancer survivors receiving chemotherapy (usually 4-5 months) at the investigators institution, for at least 8 sessions combined with at least 8 weeks of home-practice, in 25 women receiving chemotherapy for breast cancer.

ELIGIBILITY:
inclusion criteria:

* Women 20-75 years old
* Diagnosed with breast cancer
* Scheduled to begin chemotherapy at Mayo Clinic Rochester

Exclusion criteria

* Pregnant
* Practicing mindfulness

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Feasibility - percentage of patients recruited from those approached, percentage of patients who dropped off, percentage of patients who are compliant (attending more than 75% of recommended sessions) | While receiving chemotherapy (usually 4-5 months)

SECONDARY OUTCOMES:
Stress - measured by the Perceived Stress Scale - statistically and clinically significant reductions in stress | 7-8 months
  Stress will be measured before the start of chemotherapy, monthly while receiving chemotherapy (usually 4-5 months) and at 3 months after chemotherapy

OTHER OUTCOMES:
Fatigue - Multidimensional Fatigue Symptom Inventory -Short Form statistically and clinically significant reductions in fatigue score | 7-8 months
  Fatigue will be measured by the before the start of chemotherapy, monthly while receiving chemotherapy (usually 4-5 months) and at 3 months after chemotherapy
Quality of life measured by the Functional Assessment of Cancer Therapy - Breast - statistically and clinically significant improvement in quality of life | 7-8 months
  Quality of life will be measured before the start of chemotherapy, monthly while receiving chemotherapy (usually 4-5 months) and at 3 months after chemotherapy
Sleep measured by the Pittsburgh Sleep Quality Index -statistically and clinically significant improvements in sleep | 7-8 months
  Sleep will be measured before the start of chemotherapy, monthly while receiving chemotherapy (usually 4-5 months) and at 3 months after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Stan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials